CLINICAL TRIAL: NCT07344883
Title: Effects of Music on Pain in Orthopedic Patients With Distal Radius Fractures Undergoing Non-surgical Reduction: a Randomized Controlled Trial
Brief Title: Effects of Music on Procedural Pain in Distal Radius Fracture Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Massimo Guasconi, RN, PhD, Azienda Unita Sanitaria Locale di Piacenza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PolSound
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pain; Blood Pressure; Heart Rate; Music Therapy; Nursing
Keywords: nursing; musictherapy; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data processing will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1-Patient-preferred music (Experimental): After enrolment and baseline assessment (NRS, heart rate, blood pressure - T0), patients allocated to the intervention groups will receive a 20-minute music session before fracture reduction, followed by reassessment of outcomes at T1 and CRF completion.
  Group 1 will listen to patient-preferred music via headphones. Music will be administered at the patient's bedside or in the treatment area, ensuring privacy, minimal distractions, and patient comfort.
  Interventions: Other: Music intervention Group 1
- Group 2-Standardized music playlist (Experimental): After enrolment and baseline assessment (NRS, heart rate, blood pressure - T0), patients allocated to the intervention groups will receive a 20-minute music session before fracture reduction, followed by reassessment of outcomes at T1 and CRF completion.
  Group 2 will listen to a standardized music playlist selected by a music therapist (instrumental, slow tempo 60-80 BPM, stable dynamics, moderate volume).
  Music will be administered at the patient's bedside or in the treatment area, ensuring privacy, minimal distractions, and patient comfort.
  Interventions: Other: Music intervention Group 2
- Group 3- NO MUSICTHERAPY (No Intervention): The control group will receive standard care without music during the same time interval.

INTERVENTIONS:
Other: Music intervention Group 1 — After enrolment and baseline assessment (NRS, heart rate, blood pressure - T0), patients allocated to the intervention groups will receive a 20-minute music session before fracture reduction, followed by reassessment of outcomes at T1 and CRF completion.
  Group 1 will listen to patient-preferred music via headphones. Music will be administered at the patient's bedside or in the treatment area, ensuring privacy, minimal distractions, and patient comfort.
  Arms: Group 1-Patient-preferred music
Other: Music intervention Group 2 — After enrolment and baseline assessment (NRS, heart rate, blood pressure - T0), patients allocated to the intervention groups will receive a 20-minute music session before fracture reduction, followed by reassessment of outcomes at T1 and CRF completion.
  Group 2 will listen to a standardized music playlist selected by a music therapist (instrumental, slow tempo 60-80 BPM, stable dynamics, moderate volume).
  Music will be administered at the patient's bedside or in the treatment area, ensuring privacy, minimal distractions, and patient comfort.
  Arms: Group 2-Standardized music playlist

SUMMARY:
This randomized controlled trial (RCT) evaluates the effectiveness of music as a complementary intervention for pain control during non-surgical reduction of distal radius fractures in orthopedic patients. Distal radius fractures are among the most common traumatic injuries presenting to emergency departments and are frequently associated with intense procedural pain and significant physiological stress responses. Despite standard pharmacological analgesia, optimal pain management during fracture reduction remains a clinical challenge, and evidence regarding non-pharmacological adjuncts in the emergency orthopedic setting is still limited The study will enroll 192 adult patients admitted to the orthopedic emergency departments of AUSL Piacenza and AOU Parma with distal radius fractures requiring closed reduction. Participants will be randomly assigned (1:1:1) to one of three groups: a 20-minute session of patient-preferred music, a 20-minute session of standardized music selected by a music therapist, or standard care without music. Pain intensity will be assessed using the Numerical Rating Scale (NRS), while physiological stress will be evaluated through heart rate and blood pressure measurements, collected at baseline (T0) and 20 minutes later (T1), immediately after the reduction procedure The trial is designed as a prospective, randomized, controlled study with blinded data analysis, and all data will be collected and managed in compliance with current privacy and data protection regulations. By generating robust evidence on a low-cost, safe, and easily implementable intervention, the PolSound trial aims to improve procedural pain management and patient experience in emergency orthopedic care, potentially supporting the integration of music-based interventions into standard analgesic protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, 18 years of age or older
* Patients with distal radius fracture requiring non-surgical (closed) reduction
* Able to provide informed consent

Exclusion Criteria:

* Patients with severe hearing impairment
* Patients diagnosed with cognitive or psychiatric disorders
* Patients requiring emergency/urgent intervention
* Open fractures (exposed fractures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Difference in Numerical Rating Scale (NRS) pain score between T0 and T1 | Baseline and 20 minutes after baseline
  Difference in procedural pain intensity after 20 minutes compared with baseline, evaluated by NRS scores between T0 and T1.
  The NRS is an 11-point numeric scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity. A reduction in NRS score reflects improved pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- AUSL of Piacenza, Piacenza, PC, Italy

IPD SHARING:
Plan to Share IPD: Undecided